CLINICAL TRIAL: NCT06904872
Title: A Phase 2, Placebo-Controlled, Randomized, Double-Blind Study of 2 Doses of Crofelemer for the Treatment of Adult Patients With Short Bowel Syndrome and Intestinal Failure (SBS-IF) Without Colon-in-continuity (CIC)
Brief Title: Safety and Efficacy of Crofelemer in Adult Patients With Short Bowel Syndrome and Intestinal Failure (SBS-IF) Without Colon-in-continuity (CIC)
Acronym: CRO-SBS-IF
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Napo Therapeutics, S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NP303-501; 2024-511994-31-00 (EU CTIS Number)
Record Dates: First submitted 2025-03-10; First posted 2025-04-01 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Short Bowel Syndrome; Malabsorption Syndromes; Short Gut Syndrome; Post-Op Complication; Functional Gastrointestinal Disorders
Keywords: Short Bowel Syndrome
MeSH Terms: conditions — Short Bowel Syndrome; Malabsorption Syndromes; Postoperative Complications; Gastrointestinal Diseases | interventions — Solutions

STUDY DESIGN:
Intervention Model Description: Eligible patients who have met the stabilization criteria above will be randomized to one of the following treatment groups and entered into the 24-week double-blind treatment period:
  * Crofelemer 3 mg/kg/dose TID, morning, midday and evening;
  * Crofelemer 10 mg/kg/dose TID, morning, midday and evening;
  * Matched placebo TID, morning, midday and evening.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Crofelemer 3 mg/kg/dose three times daily (TID) (Experimental): Participants randomized to the Crofelemer 3 mg/kg/dose arm will receive Crofelemer 3 mg/kg/dose by oral route three times per day (TID) morning, midday, and evening for 24 weeks.
  Interventions: Drug: Crofelemer Powder for Oral Solution
- Crofelemer 10 mg/kg/dose three times daily (TID) (Experimental): Participants randomized to the Crofelemer 10 mg/kg/dose arm will receive Crofelemer 10 mg/kg/dose by oral route three times per day (TID) morning, midday, and evening for 24 weeks.
  Interventions: Drug: Crofelemer Powder for Oral Solution
- Matched Placebo three times per day (TID) (Placebo Comparator): Participants randomized to the matched placebo arm will receive matched placebo by oral route three times per day (TID) morning, midday, and evening for 24 weeks.
  Interventions: Drug: Matched Placebo Powder for Oral Solution

INTERVENTIONS:
Drug: Crofelemer Powder for Oral Solution — Crofelemer Powder for Oral Solution
  Arms: Crofelemer 10 mg/kg/dose three times daily (TID); Crofelemer 3 mg/kg/dose three times daily (TID)
Drug: Matched Placebo Powder for Oral Solution — Matched Placebo Powder for Oral Solution
  Arms: Matched Placebo three times per day (TID)

SUMMARY:
A 24-week, randomized, placebo-controlled, double-blind study to evaluate the efficacy, safety and tolerability of crofelemer in patients with Short Bowel Syndrome and Intestinal Failure (SBS-IF) without colon-in-continuity (CIC) requiring parenteral support (PS).

Blinded study drug will be administered orally (or enterally) three times daily (TID) as a novel crofelemer formulation, Crofelemer Powder for Oral Solution, or a matching placebo powder formulation for oral solution.

Patients will be randomized in a 1:1:1 ratio to crofelemer 3 mg/kg/dose TID, crofelemer 10 mg/kg/dose TID or placebo and randomization will be stratified by baseline PS volume (≤4 or >4 L/week).

DETAILED DESCRIPTION:
This is a 24-week, randomized, placebo-controlled, double-blind study to evaluate the efficacy, safety and tolerability of crofelemer in patients with Short Bowel Syndrome and Intestinal Failure (SBS-IF) without colon-in-continuity (CIC) requiring parenteral support (PS).

After an up to 4-week screening period and a PS stabilization period that will last from 2 to 12 weeks, eligible patients who have meet the stabilization requirements will be randomized 1:1:1 to the following treatment groups and entered into the 24-week double-blind treatment period:

* Crofelemer 3 mg/kg/dose TID, morning, midday and evening;
* Crofelemer 10 mg/kg/dose TID, morning, midday and evening;
* Matched placebo TID, morning, midday and evening.

Visits during the 24-week treatment period will be performed at baseline (Day 0) and after 1, 2, 4, 8, 12, 16, 20 and 24 weeks of treatments.

At the end of the 24-week treatment period, patients will be followed up for 4 weeks for safety.

For the primary and secondary objectives, changes between the two crofelemer and placebo arms will be assessed over the 24-week treatment period versus baseline.

ELIGIBILITY:
Inclusion Criteria

Patients will be enrolled in the study if they meet all the following criteria:

1. Patients must understand and provide written informed consent before they can participate in the study. They must understand the study procedures and be willing to complete the required assessments;
2. Male and female patients aged ≥ 18 years;
3. SBS patients with intestinal failure and without colon-in-continuity who are not eligible or not willing to receive an approved marketed GLP-2;
4. Patients with history of SBS resulting in intestinal failure caused by a major intestinal resection (e.g., injury, cancer*, Crohn's disease, vascular disease, volvulus) without colon-in-continuity (patients with duodenostomy, Jejunostomy or Ileostomy). Intestinal failure will be defined according to the recommendations of the European Society for Clinical Nutrition and Metabolism (ESPEN), i.e., a reduction of gut function below the minimum necessary for the absorption of macronutrients and/or water and electrolytes, such that intravenous (IV) supplementation is required to maintain health and/or growth. *Patients with history of cancer, should be in remission for the last 6 months and with not ongoing anticancer therapy (long-term hormonal therapy is allowed).
5. Minimum remaining length of 100 cm of small bowel;
6. At least 6 months elapsed since last surgical bowel resection;
7. No restorative surgery planned during the entire study period;
8. Patients with at least 4 continuous months of PS dependency (parenteral nutrition and/or intravenous fluids);
9. Chronic non-infectious diarrhoea defined as passage of at least 1 loose watery stool per day for more than 4 consecutive weeks.
10. Patients receiving stable parenteral support (fluids, electrolytes and/or nutrients) at least three days per week and a minimum of 2 liters of PS per week, to meet caloric, fluid or electrolytes needs;
11. Patients with Crohn's disease will have to be in clinical remission for ≥ 12 weeks;
12. Patients must be able to ingest solid or semi-solid foods and drink fluids;
13. If taken at screening, use of antimotility and antidiarrheal agents (loperamide, diphenoxylate, codeine and other opiates), H2-receptor antagonists, proton pump inhibitors, bile sequestering agents, oral glutamine, diuretics and oral rehydration solutions is required to be at stable average weekly doses for at least 4 weeks prior to screening evaluations;
14. If female and of child-bearing potential, the patient must use an "acceptable effective contraceptive measure" for the entire study duration and for 4 weeks after the last dose. Acceptable birth control methods that result in a failure rate of more than 1% per year include: progestogen-only oral hormonal contraception, where inhibition of ovulation is not the primary mode of action male or female condom with or without spermicide cap, diaphragm or sponge with spermicide (A combination of male condom with either cap, diaphragm or sponge with spermicide (double barrier methods) are also considered acceptable). Male patients must agree to use an acceptable form of birth control and to not donate sperm during the study and for 4 weeks after the last dose.
15. If female and child-bearing potential, the patient must have a negative urine pregnancy test prior the first administration of the investigational product;
16. Satisfactory general health status as determined by the investigator based on current medical status, medical history and physical examination.

Exclusion criteria

Patients cannot be enrolled in the study if they meet any of the following criteria:

1. Body mass index (BMI) <17.5 or >30 kg/m2;
2. Presence of clinically significant intestinal adhesions and/or chronic abdominal pain that can interfere with the conduct of the study;
3. Patients with radiological (Radiography and/or CT) signs of bowel dilatation or pseudo-obstruction;
4. Active Crohn's disease as evaluated by standard procedures employed by the investigator;
5. Inflammatory bowel disease (IBD) that required immunosuppressant therapy that has been introduced or changed within last 3 months or treatment with biologics within the last 6 months;
6. Intestinal or other major surgery scheduled within the time frame of the study;
7. Visible blood in the stool within the last 12 weeks;
8. Ongoing radiation enteritis or the presence of damaged enteral tissue due to radiation enteritis, scleroderma, celiac disease, refractory or tropical sprue;
9. Compromised immune system (e.g., acquired immune deficiency syndrome [AIDS], severe combined immunodeficiency);
10. Inadequate hepatic function: alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) and/or total bilirubin and/or alkaline phosphatases > 2 times the patient's average relative values in the last 3 months;
11. Inadequate renal function: serum creatinine or blood urea nitrogen > 2 times the Upper Normal Limit (UNL);
12. Urine sodium <20 mmol/day;
13. More than four SBS-related hospital admissions (unless one or more admissions were to rule out line sepsis) within the past 12 months or hospital admission within the last 4 weeks;
14. Concurrent or past use of infliximab, growth hormone or growth factors such as native glucagon-like peptide-2 (GLP-2) or other biological therapy within the last 12 weeks;
15. Use of systemic corticosteroids, methotrexate, cyclosporine, tacrolimus, sirolimus, octreotide, intravenous glutamine within the last 4 weeks;
16. Use of antibiotics within the last week or active infection;
17. History of alcohol abuse (Drinking more than 12 g/day of alcohol for women and 24 g/day of alcohol for men) or drug abuse within the last year;
18. Pregnant or lactating women;
19. History of psychiatric illnesses which lead to consider the patient as incapacitated and prevent him/her to provide informed consent;
20. History of any other uncontrolled chronic or acute concomitant disease which, in the Investigator's opinion, would contraindicate study participation or confound interpretation of the results;
21. Patient not capable of understanding or not willing to adhere to the study visit schedules and other protocol requirements;
22. Participation in any other interventional clinical study within five times the half-life of the investigational medicinal product / relevant metabolites (of the previous clinical study) or 4 weeks (whichever is longer) prior to screening;
23. Known hypersensitivity/allergy to any component of the IP.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-05-29 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | 24 weeks
  Frequency of Treatment-Emergent-Adverse Events
Safety and Tolerability | 24 weeks
  Frequency of IP interruption and/or discontinuation considered related to the study drug
Preliminary Efficacy | 24 weeks
  Change in weekly parenteral support (PS: parenteral nutrition (PN) and/or intravenous (IV) fluid volume) from baseline, by recording PS volume in the patient daily diary
Preliminary Efficacy | 24 weeks
  Change in weekly stool volume from baseline, by measuring and recording daily stool volume in the patient daily diary

SECONDARY OUTCOMES:
Change in parenteral support volume | 24 weeks
  Change from baseline in weekly PS volume at different study timepoints, as recorded in the patient daily diary
Change in parenteral support calories intake | 24 weeks
  Change in total number of calories administered, as detailed on the PS prescription written by the study doctor
Change in parenteral support electrolytes intake | 24 weeks
  Change in total number of electrolytes administered, as detailed on the PS prescription written by the study doctor
Change in weekly oral fluid volume intake | 24 weeks
  Change from baseline in weekly oral fluid volume intake, as recorded in the patient daily diary
Proportion of patients with change in number of days/week of PS | 24 weeks
  Proportion of patients with at least one day reduction in weekly PS
Number of days/week of PS | 24 weeks
  Change in number of days/week of PS requirements from baseline
Change in volume of loose/watery stool | 24 weeks
  Change from baseline in weekly loose/watery stools as measured by the volume in the ostomy bag or other measuring devices and recorded in the patient daily diary
Changes from baseline in stool consistency | 24 weeks
  Recording stool consistency of each stool using the 7-point Bristol Stool Scale in the patient daily diary
Changes in laboratory parameters | 24 weeks
  Changes from baseline of individual lab values within a chemistry and metabolic panel analysis
Changes in physical examination | 24 weeks
  Changes from baseline in physical examination findings (such as head, ears, eyes, nose, mouth, skin, heart, lung, lymph nodes, gastrointestinal, skeletal, and neurological signs and symptoms)

OTHER OUTCOMES:
Changes in Quality of life (QoL) | 24 weeks
  Measuring Quality of Life through administration of SBS-QoL questionnaire (17 questions to be responded with a visual analog scale) together with additional daily diary questions

CONTACTS AND LOCATIONS:
Locations (8):
- Germany (5):
  - Universitäatsklinik RWTH, Aachen
  - Charité Universitätsmedizin, Berlin
  - Universitätsklinikum, Essen
  - Asklepios Klinik St. Georg, Hamburg
  - Universitätsmedizin, Rostock
- Italy (3):
  - Azienda Ospedaliero-Universitaria di Bologna Policlinico S. Orsola-Malpighi, Bologna
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - Ospedale Università di Padova, Padua

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guillen B, Atherton NS. Short Bowel Syndrome. 2023 Jul 17. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK536935/ PMID 30725620
- [Background] Guy MK, Teixeira A, Lalani AS et al. Effects of oral on neratinib-induced diarrhea in beagle dogs. Cancer Res 2020;80(16) Supplement (Abstract#580).
- [Background] Wales PW, Christison-Lagay ER. Short bowel syndrome: epidemiology and etiology. Semin Pediatr Surg. 2010 Feb;19(1):3-9. doi: 10.1053/j.sempedsurg.2009.11.001. PMID 20123268
- [Background] Vanderhoof JA, Langnas AN. Short-bowel syndrome in children and adults. Gastroenterology. 1997 Nov;113(5):1767-78. doi: 10.1053/gast.1997.v113.pm9352883.
- [Background] Tradtrantip L, Namkung W, Verkman AS. Crofelemer, an antisecretory antidiarrheal proanthocyanidin oligomer extracted from Croton lechleri, targets two distinct intestinal chloride channels. Mol Pharmacol. 2010 Jan;77(1):69-78. doi: 10.1124/mol.109.061051. Epub 2009 Oct 6. PMID 19808995
- [Background] Thompson JS. Short Bowel Syndrome and Malabsorption - Causes and Prevention. Viszeralmedizin. 2014 Jun;30(3):174-8. doi: 10.1159/000363276. PMID 26288591
- [Background] Terrin G, Scipione A, De Curtis M. Update in pathogenesis and prospective in treatment of necrotizing enterocolitis. Biomed Res Int. 2014;2014:543765. doi: 10.1155/2014/543765. Epub 2014 Jul 17. PMID 25147804
- [Background] Tappenden KA. Pathophysiology of short bowel syndrome: considerations of resected and residual anatomy. JPEN J Parenter Enteral Nutr. 2014 May;38(1 Suppl):14S-22S. doi: 10.1177/0148607113520005. Epub 2014 Feb 5. PMID 24500909
- [Background] Schalamon J, Mayr JM, Hollwarth ME. Mortality and economics in short bowel syndrome. Best Pract Res Clin Gastroenterol. 2003 Dec;17(6):931-42. doi: 10.1016/s1521-6918(03)00079-9. PMID 14642858
- [Background] Pironi L, Arends J, Bozzetti F, Cuerda C, Gillanders L, Jeppesen PB, Joly F, Kelly D, Lal S, Staun M, Szczepanek K, Van Gossum A, Wanten G, Schneider SM; Home Artificial Nutrition & Chronic Intestinal Failure Special Interest Group of ESPEN. ESPEN guidelines on chronic intestinal failure in adults. Clin Nutr. 2016 Apr;35(2):247-307. doi: 10.1016/j.clnu.2016.01.020. Epub 2016 Feb 8. PMID 26944585
- [Background] Parrish CR, DiBaise JK. Managing the Adult Patient With Short Bowel Syndrome. Gastroenterol Hepatol (N Y). 2017 Oct;13(10):600-608. PMID 29230136
- [Background] Nee J, Salley K, Ludwig AG, Sommers T, Ballou S, Takazawa E, Duehren S, Singh P, Iturrino J, Katon J, Lee HN, Rangan V, Lembo AJ. Randomized Clinical Trial: Crofelemer Treatment in Women With Diarrhea-Predominant Irritable Bowel Syndrome. Clin Transl Gastroenterol. 2019 Dec;10(12):e00110. doi: 10.14309/ctg.0000000000000110. PMID 31800542
- [Background] Mangel AW, Chaturvedi P. Evaluation of crofelemer in the treatment of diarrhea-predominant irritable bowel syndrome patients. Digestion. 2008;78(4):180-6. doi: 10.1159/000185719. Epub 2008 Dec 18. PMID 19092244
- [Background] Lochs H, Dejong C, Hammarqvist F, Hebuterne X, Leon-Sanz M, Schutz T, van Gemert W, van Gossum A, Valentini L; DGEM (German Society for Nutritional Medicine); Lubke H, Bischoff S, Engelmann N, Thul P; ESPEN (European Society for Parenteral and Enteral Nutrition). ESPEN Guidelines on Enteral Nutrition: Gastroenterology. Clin Nutr. 2006 Apr;25(2):260-74. doi: 10.1016/j.clnu.2006.01.007. Epub 2006 May 15. PMID 16698129
- [Background] Kumpf VJ. Pharmacologic management of diarrhea in patients with short bowel syndrome. JPEN J Parenter Enteral Nutr. 2014 May;38(1 Suppl):38S-44S. doi: 10.1177/0148607113520618. Epub 2014 Jan 24. PMID 24463352
- [Background] Jeppesen PB. Spectrum of short bowel syndrome in adults: intestinal insufficiency to intestinal failure. JPEN J Parenter Enteral Nutr. 2014 May;38(1 Suppl):8S-13S. doi: 10.1177/0148607114520994. Epub 2014 Jan 31. PMID 24486858
- [Background] Jeppesen PB. Teduglutide, a novel glucagon-like peptide 2 analog, in the treatment of patients with short bowel syndrome. Therap Adv Gastroenterol. 2012 May;5(3):159-71. doi: 10.1177/1756283X11436318. PMID 22570676
- [Background] Jeppesen PB, Pertkiewicz M, Messing B, Iyer K, Seidner DL, O'keefe SJ, Forbes A, Heinze H, Joelsson B. Teduglutide reduces need for parenteral support among patients with short bowel syndrome with intestinal failure. Gastroenterology. 2012 Dec;143(6):1473-1481.e3. doi: 10.1053/j.gastro.2012.09.007. Epub 2012 Sep 11. PMID 22982184
- [Background] Jeppesen PB, Gilroy R, Pertkiewicz M, Allard JP, Messing B, O'Keefe SJ. Randomised placebo-controlled trial of teduglutide in reducing parenteral nutrition and/or intravenous fluid requirements in patients with short bowel syndrome. Gut. 2011 Jul;60(7):902-14. doi: 10.1136/gut.2010.218271. Epub 2011 Feb 11. PMID 21317170
- [Background] Janssen MF, Pickard AS, Golicki D, Gudex C, Niewada M, Scalone L, Swinburn P, Busschbach J. Measurement properties of the EQ-5D-5L compared to the EQ-5D-3L across eight patient groups: a multi-country study. Qual Life Res. 2013 Sep;22(7):1717-27. doi: 10.1007/s11136-012-0322-4. Epub 2012 Nov 25. PMID 23184421
- [Background] Holodniy M, Koch J, Mistal M, Schmidt JM, Khandwala A, Pennington JE, Porter SB. A double blind, randomized, placebo-controlled phase II study to assess the safety and efficacy of orally administered SP-303 for the symptomatic treatment of diarrhea in patients with AIDS. Am J Gastroenterol. 1999 Nov;94(11):3267-73. doi: 10.1111/j.1572-0241.1999.01535.x. PMID 10566728
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] Gabriel SE, Davenport SE, Steagall RJ, Vimal V, Carlson T, Rozhon EJ. A novel plant-derived inhibitor of cAMP-mediated fluid and chloride secretion. Am J Physiol. 1999 Jan;276(1):G58-63. doi: 10.1152/ajpgi.1999.276.1.G58. PMID 9886979
- [Background] Capriati T, Mosca A, Alterio T, Spagnuolo MI, Gandullia P, Lezo A, Lionetti P, D'Antiga L, Fusaro F, Diamanti A. To Wean or Not to Wean: The Role of Autologous Reconstructive Surgery in the Natural History of Pediatric Short Bowel Syndrome on Behalf of Italian Society for Gastroenterology, Hepatology and Nutrition (SIGENP). Nutrients. 2020 Jul 18;12(7):2136. doi: 10.3390/nu12072136. PMID 32708377
- [Background] Camilleri M. Intestinal secretory mechanisms in irritable bowel syndrome-diarrhea. Clin Gastroenterol Hepatol. 2015 Jun;13(6):1051-7; quiz e61-2. doi: 10.1016/j.cgh.2014.07.020. Epub 2014 Jul 17. PMID 25041862
- [Background] Cagir B. Short Bowel Syndrome. Clinical Presentation. emedicine Medscape 2017.
- [Background] Braga M, Ljungqvist O, Soeters P, Fearon K, Weimann A, Bozzetti F; ESPEN. ESPEN Guidelines on Parenteral Nutrition: surgery. Clin Nutr. 2009 Aug;28(4):378-86. doi: 10.1016/j.clnu.2009.04.002. Epub 2009 May 21. PMID 19464088
- [Background] Berghofer P, Fragkos KC, Baxter JP, Forbes A, Joly F, Heinze H, Loth S, Pertkiewicz M, Messing B, Jeppesen PB. Development and validation of the disease-specific Short Bowel Syndrome-Quality of Life (SBS-QoL) scale. Clin Nutr. 2013 Oct;32(5):789-96. doi: 10.1016/j.clnu.2012.12.001. Epub 2012 Dec 12. PMID 23274148